CLINICAL TRIAL: NCT04341610
Title: Allogeneic Adipose Tissue Derived Mesenchymal Stromal Cell Therapy for Treating Patients With Severe Respiratory COVID-19. A Danish, Double-blind, Randomized Placebo-controlled Study
Brief Title: ASC Therapy for Patients With Severe Respiratory COVID-19
Acronym: ASC COVID-19
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not approved by ethical committee
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, JKastrup, Professor MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT number: 2020-001330-36
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Tract Diseases
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Intervention Model Description: Double-blind placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASC (Active Comparator): 100 million allogeneic adipose-derived mesenchymal stromal cell
  Interventions: Drug: Stem Cell Product
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Stem Cell Product

INTERVENTIONS:
Drug: Stem Cell Product — 100 million allogeneic adipose-derived mesenchymal stromal cells diluted in 100 ml saline

SUMMARY:
The emerging field of stem cell therapy holds promise of treating a variety of diseases. Especially the mesenchymal stromal cells from bone marrow or adipose tissue (ASCs) have proven their potential for regenerative therapy in patients with ischemic heart disease. Both of these cell types have putative immunomodulatory properties, as they have demonstrated their ability to evade recognition and actively suppress the immune system.

This knowledge is transferred into studies with COVID-19 patients having severe pulmonary dysfunction, to modify the virus induced immunological and inflammatory activity involved in the progression of disease often leading to prolonged ICU stay and in some occasion's death.

We will conduct a clinical trial in which patients with COVID-19 and severe pulmonary symptoms will be randomized to either placebo or treatment with allogeneic CSCC_ASCs from adipose tissue. The aim is to assess the impact of CSCC_ASCs on the activated immune system and clinical efficacy on pulmonary function.

The perspective is that this new information can be of pivotal importance and potentially be a paradigm shift for the clinical problems and severe outcome seen in some patients with severe COVID-19 and other severe diseases with Acute Respiratory Distress Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-80 years
* Confirmed HCoV-19 infection
* Temperature above 38.0o C
* Pulmonary symptoms and signs, at least one of the following before clinical decision for intubation and respirator treatment:

  1. Respiratory distress, RR ≥ 30/min;
  2. Oxygen saturation ≤ 93% at rest state;
  3. Arterial partial pressure of oxygen (PaO2) / Fraction of inspiration O2 (FiO2) ≤ 300mmHg, 1mmHg=0.133kPa
* Pneumonia that is judged by chest radiograph or computed tomography
* In respirator and possible for treatment within the first 24 hours

Exclusion Criteria:

* Patients that have need for additional immunosuppressive treatment
* Patients with any past (within the past 3-5 years) or present malignancy (other than excised basal cell carcinoma).
* Co-Infection with other infectious agent.
* Females capable of becoming pregnant must have a negative pregnancy test prior to treatment. After inclusion, they must use contraceptives for 2 months following the given stem cell treatment. The pill, spiral, depot injection of progesterone, sub-dermal implantation, hormonal vaginal ring and transdermal patch regarded as safe contraceptives.
* Patients who are participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in clinical critical treatment index | day 7 from randomization

SECONDARY OUTCOMES:
Days of respirator treatment | 3 months
Improvement of clinical symptoms including duration of fever and respiratory need | 3 months
Mortality | 3 months
Marker of Immunological function -CD4+ and CD8+ T cell count | 3 months
C-reactive protein and leucocyte | 3 months
Cytokine profile | 3 months
Glomerular Filtration Rate | 3 months
Duration of hospitalization | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- 2014 Department of Cardiology, The Heart Centre, University Hospital Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided